CLINICAL TRIAL: NCT05611645
Title: A Randomized Phase II Trial of Concurrent Low-dose Bevacizumab and HSRT Versus Bevacizumab Alone for Glioblastoma at First Recurrence: HSCK-005
Brief Title: Low-dose Bevacizumab With HSRT vs BVZ Alone for GBM at First Recurrence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yun Guan, Physician, CyberKnife Center, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-798
Record Dates: First submitted 2022-10-28; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Glioma; Recurrent Glioma
MeSH Terms: conditions — Glioma | interventions — Radiosurgery; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HSRT+Low-dose Bevacizumab (Experimental): HSRT with low-dose bevacizumab every 2 weeks
  Interventions: Radiation: Hypofractionated Stereotactic Radiotherapy; Drug: Bevacizumab
- Bevacizumab (Active Comparator): Bevacizumab every 2 weeks
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Radiotherapy — Starting with low-dose bevacizumab, 25Gy in 5 fractions of 5 Gy each delivered on consecutive treatment days.
  Other Names: Hypofractionated Stereotactic Radiosurgery; Image-Guided Radiation Treatment (IGRT); Stereotactic Radiosurgery (SRS)
  Arms: HSRT+Low-dose Bevacizumab
Drug: Bevacizumab — Staring within 2 weeks of randomization, IV 5mg/kg (experimental group) or 10mg/kg (comparison group) every two weeks until disease progression.
  Other Names: anti-VEGF monoclonal antibody; rhuMAb VEGF; Avastin

SUMMARY:
This randomized phase II trial studies how well lose dose bevacizumab with Hypofractionated Stereotactic Radiotherapy (HSRT) works versus bevacizumab alone in treating patients with glioblastoma at first recurrence. The primary endpoint is 6-month progress-free survivaloverall survival after the treatment. Secondary endpoints included overall survival, objective response rate, cognitive function, quality of life and toxicity.

DETAILED DESCRIPTION:
To establish an improvement in 6-month pfs in recurrent glioblastoma patients receiving low-dose bevacizumab and re-irradiation compared with patients receiving bevacizumab alone.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age;
* Karnofsky performance status (KPS) ≥ 60;
* Original histopathologically proven diagnosis World Health Organization (WHO) Grade 3/4 glioma;
* Underwent surgery, chemoradiotherapy and adjuvant chemotherapy (Stupp Protocol) after initial diagnosis, recurrent based on the Response Assessment in Neuro-Oncology (RANO) criteria and/or histopathologically proven;
* Measurable disease;
* Estimated survival of at least 3 months, maximal diameter on T1+C MRI ≤ 3.5 cm;
* Hgb > 9 gm; absolute neutrophil count (ANC) > 1500/μl; platelets > 100,000; Creatinine < 1.5 times the upper limit of laboratory normal value; Bilirubin < 2 times the upper limit of laboratory normal value; serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) < 3 times the upper limit of laboratory normal value;
* Signed informed consent form;
* Agreed to participate the follow-up.

Exclusion Criteria:

* Prior invasive malignancy unless disease free;
* Received re-irradiation;
* More than 3 relapses or evidence of subtentorial recurrent disease or tumor greater than 6 cm in maximum diameter;
* Prior therapy with an inhibitor of vascular endothelial growth factor (VEGF) or VEGFR;
* Pregnancy or or nursing mothers;
* Participated in other trials after diagnosis of recurrent;
* Influence factors toward oral medications;
* Patients with CTCAE5.0 grade 3+ bleeding;
* Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
* Long-term unhealed wounds or fractures;
* History of organ transplantation;
* Serious diseases that endanger patients' safety or affect patients' completion of research,according to the researchers' judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival rate at 6 Months | From randomization to six months
  Prgression was defined using Response Assessment in Neuro-Oncology (RANO) Criteria. Progression-free at 6 months means patient alive without progression at 6 months. Survival rates are estimated by the Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall Survival | From randomization to last follow-up, up to approximately 24 months
  Survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Survival rates are estimated by the Kaplan-Meier method.
Progression-free Survival | From randomization to last follow-up, up to approximately 24 months
  Prgression was defined using Response Assessment in Neuro-Oncology (RANO) Criteria. Progression-free survival time is defined as time from randomization to the date of first progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method.
Objective response rate | Bimonthly up to intolerance the toxicity or progressive disease (PD), up to approximately 24 months
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Assessment in Neuro-Oncology (RANO) prior to progression or any further therapy.
Number of Participants With Grade 3+ Toxicity rate | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade refers to the severity of the AE. Estimated using an exact binomial distribution together with 95% confidence interval. The difference between the two groups will be tested using a chi square test.
Quality of Life score (QoL) | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  EORTC QLQ-C30 (version 3.0) questionnaire to evaluate the quality of life. All scales range in score from 0 to 100. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Cognitive function | Bimonthly up to intolerance the toxicity or PD, up to approximately 24 months
  Mini-Mental State Exam (MMSE, score range 0 to 30) to evaluate the cognitive function. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- CyberKnife Center, Department of Neurosurgery, Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan Y, Li J, Gong X, Zhu H, Li C, Mei G, Liu X, Pan L, Dai J, Wang Y, Wang E, Liu Y, Wang X. Safety and Efficacy of Hypofractionated Stereotactic Radiotherapy with Anlotinib Targeted Therapy for Glioblastoma at the First Recurrence: A Preliminary Report. Brain Sci. 2022 Apr 2;12(4):471. doi: 10.3390/brainsci12040471. PMID 35448002
- [Background] Guan Y, Xiong J, Pan M, Shi W, Li J, Zhu H, Gong X, Li C, Mei G, Liu X, Pan L, Dai J, Wang Y, Wang E, Wang X. Safety and efficacy of Hypofractionated stereotactic radiosurgery for high-grade Gliomas at first recurrence: a single-center experience. BMC Cancer. 2021 Feb 5;21(1):123. doi: 10.1186/s12885-021-07856-y. PMID 33546642